CLINICAL TRIAL: NCT02115061
Title: Gastric Varices Treatment: Coil + Cyanoacrylate Versus Cyanoacrylate
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 02621613100000068
Record Dates: First submitted 2014-04-03; First posted 2014-04-15 (Estimated); Last update posted 2014-04-15 (Estimated); Status verified 2012-08

CONDITIONS: Gastric Varices
Keywords: Gastric varices,coil,cyanoacrylate,treating gastric varices.
MeSH Terms: conditions — Esophageal and Gastric Varices

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cyanoacrylate (Active Comparator): This group owned fourteen patients who met all the inclusion criteria. These will be treated with cyanoacrylate.
  Treatment: cyanoacrylate
  Interventions: Device: Treatment: cyanoacrylate
- Coil + cyanocrylate (Sham Comparator): This group had fourteen patients who met all inclusion criteria. These will be treated with coil + cyanoacrylate.
  Treatment: coil + cyanoacrylate
  Interventions: Device: Treatment: coil + cyanoacrylate

INTERVENTIONS:
Device: Treatment: coil + cyanoacrylate — This group had fourteen patients who met all inclusion criteria. These will be treated with coil + cyanoacrylate.
  Other Names: Coil + cyanoacrylate
  Arms: Coil + cyanocrylate
Device: Treatment: cyanoacrylate — This group owned fourteen patients who met all the inclusion criteria. These will be treated with cyanoacrylate.
  Other Names: Cyanoacrylate
  Arms: Cyanoacrylate

SUMMARY:
The purpose of the spring is to maintain the cyanoacrylate polymer of the gastric varix, forming a conglomerate spring-cyanoacrylate, and thus preventing their migration to the adhesive embolism.

The introduction of the spring is held by a echo-guided puncture. The window can be puncture through the distal esophagus or directly in the gastric varix via retroflexion to the fundus. Another advantage of this technique is its use in the presence of bleeding, when large amounts of blood in the stomach hinders the injection of the cyanoacrylate, by pricking the distal esophagus that difficulty decreases. The first study of this technique was performed by Binmoeller et al (21) and had good results with 100% hemostasis and low rebleeding rate (16%), but more studies are needed to prove the safety and efficacy of this technique.

DETAILED DESCRIPTION:
OBJECTIVE Compare the results of the treatment of gastric varices, coil associated with cianoarilato versus cyanoacrylate in patients with systemic shunts in relation to efficacy and embolic complications.

PATIENTS, MATERIALS AND METHODS Drawing

This is a prospective clinical trial, double-blind, comparative, randomized, single center, performed on quaternary level hospital involving patients with portal hypertension with gastric varices type 2 GOV or IGV 1.

28 cirrhotic patients will be randomized to the treatment of gastric varices type GOV2 IGV1 or more cyanoacrylate Cyanoacrylate or only patients with splenorenal shunt or gastrorenal spring.

After signing the consent form, patients will undergo CT angiography to evaluate the presence of shunt and classification of the same. Patients without shunt will be excluded from the protocol.

Dopller colored portal system will also be conducted in all patients prior to treatment for analysis of portal flow.

After confirming the presence of shunt patients will be examined by echo-endoscopy for completion of treatment The following data will be collected: demographic data (age and gender), etiology of cirrhosis, degree of liver function, primary or secondary prophylaxis diameter of gastric varix, varices of the esophagus with or without signs of red color, size and type of shunt detected by CT, amount of springs inserted, number of ampoules of Cyanoacrylate injected complications (bleeding, damage to the endoscope by cyanoacrylate)

ELIGIBILITY:
Inclusion Criteria:

* Patients with portal hypertension and pseudo-tumor gastric varices type IGV1 or GOV2 and presence of gastrorenal or splenorenal shunt.

Exclusion Criteria:

* Refusal of the patient or their legal guardian.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2013-08; Primary Completion 2014-08 (Estimated); Study Completion 2014-10 (Estimated)

PRIMARY OUTCOMES:
Compare the results of the treatment of gastric varices, gastric varices treatment coil and cyanocrylate versus cyanocrylate in 28 patients with systemic shunts in relation to efficacy and embolic complications. | Four months after patient recruitment.
  Patient recruitment, the signing of the terms and data collection will be carried out between September 2012 and August 2014. Data analysis and statistical studies between September and October 2014. The scheduled date for completion of the study is the December 2014.
  The monitoring will be performed with endoscopy and endoscopic ultrasound at 1, 4 and 10 months after the procedure. Analyzed the recurrence and clinical outcome, with completion of new questionnaires.

CONTACTS AND LOCATIONS:
Overall Officials: Maíra R de Almeida, Study Chair — Hospital das Clínicas da FMUSP; Dalton Chaves, Principal Investigator — Hospital das Clínicas FMUSP
Locations (1):
- Hospital das Clínicas da FMUSP, São Paulo, São Paulo, Brazil